CLINICAL TRIAL: NCT01638429
Title: Methane Production and Glycemic Regulation in Pre-diabetic Subjects: Role of Methane in Glycemic Control
Brief Title: Role of Methane in Glycemic Control
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Ruchi Mathur, Director, Clinical Diabetes Outpatient Treatment and Education Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25182
Record Dates: First submitted 2012-04-30; First posted 2012-07-11 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-01

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Neomycin; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obese/overweight, prediabetic methane positive (Experimental): Neomycin Rifaximin
  Interventions: Drug: Neomycin; Drug: Rifaximin

INTERVENTIONS:
Drug: Neomycin — Neomycin: 500mg po bid for 10 days
Drug: Rifaximin — Rifaximin: 550mg po tid for 10 days

SUMMARY:
The purpose of this study is to determine how certain types of bacteria in the human gut may affect weight gain, and contribute to the development of diabetes.

The investigators initial studies have shown that gut bacteria that produce methane may directly affect weight gain. These bacteria, called methanogens, produce methane gas as a byproduct, which can be detected through breath testing. Methane can slow the passage of food through the intestines, which would allow extra time for uptake and absorption of nutrients and calories, and might contribute to weight gain. The investigators have also found that people who have increased levels of methane-producing bacteria in their intestines also have higher levels of glucose in their blood. Therefore, control of how the body responds to insulin and uses glucose may be altered in methane-producing individuals.

This research study is designed to test the investigational use of the drugs neomycin and rifaximin that have been approved by the U.S Food and Drug Administration (FDA). While neomycin is FDA-approved for treating skin infections, preparing the bowel for surgery, and hepatic encephalopathy (a condition that occurs when a damaged liver cannot remove the toxins that a healthy liver normally would), and rifaximin is FDA-approved for treating travelers' diarrhea, they are not yet approved to be used together for the treatment of methanogens or obesity.

DETAILED DESCRIPTION:
Pre-diabetes is defined by impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) and affects more than 40% of US adults. While glycemic dysregulation and insulin resistance are central to the progression from pre-diabetes to diabetes, obesity also plays a key role. Research has begun to define the relationship between gut flora, metabolism and weight gain. Animal studies have linked a specific methanogen, Methanobrevibacter smithii, to weight gain, and in humans we have found that increased methane on breath test is associated both with increased body mass index (BMI) and higher blood glucose levels. We also found that methane gas directly slows gut transit by 59% in an in vivo animal model. We hypothesize that this slowing of transit could result in a greater time to harvest nutrients and absorb calories, representing a potential mechanism for elevated post-prandial glycemic excursions and weight gain. In this study, we will test this hypothesis by determining the effects of enteric methane production on glucose excursions, gut transit and energy utilization in obese or overweight, prediabetic, adult subjects.

We will explore the relationship between methane, M. smithii, obesity and gut transit in human subjects using objective measures of metabolic function, glucose excursions, energy utilization and transit studies, to evaluate whether intestinal methane production is associated with a higher incidence of diabetes risk in an obese study population. We will then repeat testing following a course of antibiotics known to eliminate methanogens. This will potentially provide novel therapies for the pre-diabetic patient, and allow new avenues for research.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old with pre-diabetes (hemoglobin a1c of 5.7-6.4%)
* BMI > 25.0
* presence of methane on a breath sample (>3ppm)

Exclusion Criteria:

Subjects will be excluded from the study if they exhibit any of the following:

* Diabetes/diabetes medications
* Prokinetic medication
* Pregnancy
* History of bariatric or intestinal surgery (other than cholecystectomy or appendectomy)
* Unstable thyroid disease
* An active weight loss treatment/plan
* Smoking
* Dietary restrictions (lactose intolerance, vegan etc)
* Other inability to comply with the study procedures, including known allergy to the study antibiotics (neomycin and rifaximin)
* Active inflammatory bowel disease (celiac, Crohn's disease, ulcerative colitis)
* Antibiotic use in the past month
* Subjects who do not have a microwave (for reheating study meals) and a freezer (for storing leftovers and stool samples) will be excluded from this study.
* Subjects who have an aspirin sensitivity
* Proton pump inhibitor medications or antacids
* History of bezoar
* Disorders of swallowing
* Suspected strictures, fistulas or physiological GI obstruction
* GI surgery within 3 months
* Severe dysphagia to food or pills
* Diverticulitis
* Subjects who use an implanted or portable electromechanical device such as a cardiac pacemaker or infusion pump
* Subject who have a peanut allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruchi Mathur, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open for recruitment from April 12, 2012 - Dec 31, 2013 Setting: Tertiary care center
Pre-assignment Details: A total of 12 subjects were consented to participate. 1 subject withdrew prior to completing the study.
Groups:
- Obese/Overweight, Prediabetic Methane Positive Subjects: Neomycin Rifaximin
  Neomycin: Neomycin: 500mg po bid for 10 days
  Rifaximin: Rifaximin: 550mg po tid for 10 days
Period: Overall Study
Arm/Group | Obese/Overweight, Prediabetic Methane Positive Subjects
Started | 12
Pre-treatment Testing | 11
Antibiotic Treatment | 11
Post-treatment Testing | 11
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Obese/Overweight, Prediabetic Methane Positive Subjects
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.17 (7.71)
A1c (%) [Mean (Standard Deviation); unit: Percent] | 5.72 (0.60)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Eradicated Methane on Breath Test
Description: Number of subjects who exhibited a decrease in breath methane levels to below detectable (below 3ppm) following antibiotic treatment.
  After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics. Post-treatment breath tests were performed within 2 weeks (14 days) of completing the course of antibiotics.
Time Frame: Baseline and 1-14 days following completion of antibiotic treatment
Measure: Number; unit: participants
Arm/Group | Obese/Overweight, Prediabetic Methane Positive
Number analyzed (Participants) | 11
participants | 8

2. Primary Outcome: Stool Methanogen Levels
Description: Stool methanogen levels were measured in all subjects before and after antibiotic treatment. After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics. Post-treatment stool samples were collected within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days.
  For analysis, subjects were grouped into two groups:
  Group 1 - Methane Eradicators (subjects who eradicated methane on breath test following antibiotic treatment) (N=8) Group 2 - Methane Non-eradicators (subjects who did not eradicate methane on breath test following antibiotic treatment) (N=3)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: colony forming units
Groups:
- Methane Eradicators: Subjects who eradicated methane on breath test following antibiotic treatment
- Methane Non-Eradicators: Subjects who did not eradicate methane on breath test following antibiotic treatment
Arm/Group | Methane Eradicators | Methane Non-Eradicators
Number analyzed (Participants) | 8 | 3
colony forming units
  Pre-treatment | 3.6*10^7 (9.2*10^7) | 6.86*10^8 (4.9*10^3)
  Post-treatment | 1.1*10^5 (1.3*10^5) | 9.4*10^7 (7.9*10^7)
Statistical Analysis 1: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

3. Primary Outcome: Stool Total Bacteria Levels
Description: Stool total bacteria levels were measured in all subjects before and after antibiotic treatment. After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics.Post-treatment stool samples were collected within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days. For analysis, subjects were grouped into two groups:
  Group 1 - Methane Eradicators (subjects who eradicated methane on breath test following antibiotic treatment) (N=8) Group 2 - Methane Non-eradicators (subjects who did not eradicate methane on breath test following antibiotic treatment) (N=3)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: colony forming units
Arm/Group | Methane Eradicators | Methane Non-Eradicators
Number analyzed (Participants) | 8 | 3
colony forming units
  Pre-treatment | 1.1*10^9 (7.4*10^8) | 3.7*10^8 (6.4*10^8)
  Post-treatment | 1.2*10^9 (6.3*10^8) | 8.5*10^9 (1.4*10^10)

4. Primary Outcome: Low Density Lipoprotein (LDL) Levels Before and After Antibiotic Therapy
Description: LDL levels were measured in all subjects before and after antibiotic treatment. After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics. Post-treatment blood samples were collected within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days.
  For analysis, subjects were grouped into two groups:
  Group 1 - Methane Eradicators (subjects who eradicated methane on breath test following antibiotic treatment) (N=8) Group 2 - Methane Non-eradicators (subjects who did not eradicate methane on breath test following antibiotic treatment) (N=3)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Methane Eradicators | Methane Non-Eradicators
Number analyzed (Participants) | 8 | 3
mg/dL
  Pre-treatment | 116 (42) | 96 (41)
  Post-treatment | 104 (46) | 111 (51)
Statistical Analysis 1: Comparison: Methane Eradicators vs Methane Non-Eradicators; P-value is comparing change in methane eradiacators before and after treatment to change in methane non-eradiacators before and after treatment; Test type: Superiority or Other; p = 0.028, t-test, 2 sided

5. Primary Outcome: Total Cholesterol Levels Before and After Antibiotic Therapy
Description: Total cholesterol levels were measured in all subjects before and after antibiotic treatment. After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics.Post-treatment blood samples were collected within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days.
  For analysis, subjects were grouped into two groups:
  Group 1 - Methane Eradicators (subjects who eradicated methane on breath test following antibiotic treatment) (N=8) Group 2 - Methane Non-eradicators (subjects who did not eradicate methane on breath test following antibiotic treatment) (N=3)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Methane Eradicators | Methane Non-Eradicators
Number analyzed (Participants) | 8 | 3
mg/dL
  Pre-treatment | 192 (51) | 173 (41)
  Post-treatment | 177 (52) | 188 (49)
Statistical Analysis 1: Comparison: Methane Eradicators vs Methane Non-Eradicators; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

6. Primary Outcome: Average Daily Caloric Loss in Stool
Description: The daily caloric loss in stool for each subject was calculated by expressing the total number of kcalories lost in stool over a 3-day period as a percentage of the total number of kcalories ingested over the same 3 days (the number of calories ingested = the number available in meals provided less the number remaining in leftovers). Caloric content for meals, leftovers, and stool was determined by bomb calorimetry. This average daily caloric loss for each group was then compared before and after antibiotic therapy.
  Post-treatment caloric harvest studies were performed within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days. For analysis, subjects were grouped into two groups:
  Group 1 - Total study population (methane eradicators and non-eradicators, N=11) Group 2 - Methane eradicators (subjects who eradicated methane on breath test following antibiotic treatment, N=8)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: %kcal lost
Groups:
- Total Study Population: All subjects (methane eradicators and non-eradicators)
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
%kcal lost
  Pre-treatment | 8.1 (2.7) | 8.3 (1.8)
  Post-treatment | 8.3 (3.8) | 8.3 (3.8)
Statistical Analysis 1: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.97, t-test, 2 sided
Statistical Analysis 2: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.85, t-test, 2 sided

7. Primary Outcome: Gastric Emptying
Description: Gastric Emptying times (minutes) were determined in all subjects before and after antibiotic treatment. After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics. Post-treatment gastric emptying studies were performed within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days. For analysis, subjects were grouped into two groups:
  Group 1 - Total study population (methane eradicators and non-eradicators, N=11) Group 2 - Methane eradicators (subjects who eradicated methane on breath test following antibiotic treatment, N=8)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
minutes
  Pre-treatment | 182.3 (72.8) | 174.9 (71.1)
  Post-treatment | 163.5 (46.8) | 164.9 (45.8)
Statistical Analysis 1: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.61, t-test, 2 sided
Statistical Analysis 2: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.45, t-test, 2 sided

8. Secondary Outcome: Bowel Symptoms - Bloating
Description: Bowel symptom scores on a visual analog scale (VAS) were compared in all subjects before and after antibiotic treatment. Scale values were from 0 to 100, where 0 indicates no symptom and 100 indicates severe symptoms.
  After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics. Post-treatment symptom scores were obtained within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days. For analysis, subjects were grouped into two groups:
  Group 1 - Total study population (methane eradicators and non-eradicators, N=11) Group 2 - Methane eradicators (subjects who eradicated methane on breath test following antibiotic treatment, N=8)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: 0-100mm visual analogue scale
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
0-100mm visual analogue scale
  Pre-treatment | 55.09 (34.18) | 66.8 (32.4)
  Post-treatment | 39.91 (33.27) | 38.9 (36.1)
Statistical Analysis 1: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.018, t-test, 2 sided
Statistical Analysis 2: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.14, t-test, 2 sided

9. Secondary Outcome: Bowel Symptoms - Abdominal Pain
Description: as for outcome 8
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: 0-100mm visual analogue scale
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
0-100mm visual analogue scale
  Pre-treatment | 23.36 (27.18) | 28.6 (30.3)
  Post-treatment | 18.18 (29.91) | 21.6 (34.7)
Statistical Analysis 1: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.43, t-test, 2 sided
Statistical Analysis 2: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.44, t-test, 2 sided

10. Secondary Outcome: Bowel Symptoms - Constipation
Description: as for outcome 8
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: 0-100mm visual analogue scale
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
0-100mm visual analogue scale
  Pre-treatment | 30.18 (29.75) | 31.0 (30.5)
  Post-treatment | 20.55 (33.90) | 22.3 (39.6)
Statistical Analysis 1: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.13, t-test, 2 sided
Statistical Analysis 2: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.25, t-test, 2 sided

11. Secondary Outcome: Bowel Symptoms - Diarrhea
Description: as for outcome 8
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: 0-100mm visual analogue scale
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
0-100mm visual analogue scale
  Pre-treatment | 23.73 (30.16) | 30.5 (32.9)
  Post-treatment | 14.64 (31.01) | 17.3 (36.0)
Statistical Analysis 1: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.29, t-test, 2 sided
Statistical Analysis 2: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.27, t-test, 2 sided

12. Secondary Outcome: Bowel Symptoms - Straining
Description: as for outcome 8
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: 0-100mm visual analogue scale
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
0-100mm visual analogue scale
  Pre-treatment | 31.64 (29.25) | 37.5 (31.8)
  Post-treatment | 21.55 (30.19) | 18.4 (34.5)
Statistical Analysis 1: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.22, t-test, 2 sided
Statistical Analysis 2: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.059, t-test, 2 sided

13. Secondary Outcome: % Stool Dry Weight
Description: % stool dry weight [total stool dry weight (g)/total stool fresh weight (g)] was determined in all subjects before and after antibiotic treatment. After baseline (pre-treatment) testing, subjects underwent a 10-day course of antibiotics. Post-treatment stool samples were obtained within 31 days (1 month) of completing the course of antibiotics. One subject received an exemption from this requirement and completed testing within 60 days. For analysis, subjects were grouped into two groups: Group 1 - Total study population (methane eradicators and non-eradicators, N=11) Group 2 - Methane eradicators (subjects who eradicated methane on breath test following antibiotic treatment, N=8)
Time Frame: Baseline and 1-60 days following completion of antibiotic treatment
Measure: Mean (Standard Deviation); unit: % stool dry weight
Arm/Group | Total Study Population | Methane Eradicators
Number analyzed (Participants) | 11 | 8
% stool dry weight
  Pre-treatment | 24.1 (5.3) | 25.1 (4.7)
  Post-treatment | 22.9 (4.4) | 22.6 (4.4)
Statistical Analysis 1: Comparison: Total Study Population; Values compared in total study population pre- and post-treatment; Test type: Superiority or Other; p = 0.33, t-test, 2 sided
Statistical Analysis 2: Comparison: Methane Eradicators; Values compared in methane eradicators only pre- and post-treatment; Test type: Superiority or Other; p = 0.075, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Obese/Overweight, Prediabetic Methane Positive Subjects
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese/Overweight, Prediabetic Methane Positive Subjects (N=11)
Loose stool (Gastrointestinal disorders) | 2 (2) — 2 subjects reported looser stools than normal after taking the study antibiotics. Loose stool is a known potential side effect of the antibiotics used in the study. Stool cutures were performed and were negative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No